CLINICAL TRIAL: NCT04899362
Title: The Impact of Serial Remote Ischemic Conditioning on Dynamic Cerebral Autoregulation in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRIC-CA
Record Dates: First submitted 2021-05-10; First posted 2021-05-24 (Actual); Results first posted 2023-12-07 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2021-05

CONDITIONS: Remote Ischemic Conditioning
Keywords: Remote Ischemic Conditioning; Dynamic Cerebral Autoregulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RIC group (Experimental): RIC was induced by 4 cycles of extremities ischemia (5-minute blood-pressure cuff inflation to 200 mm Hg, followed by 5-minute cuff deflation).All subjects will take 14 RIC intervention, blood collection and 10 dCA measurements.
  Interventions: Device: BB-RIC-D1/LAPUL Medical Devices Co, Ltd, China; Procedure: Intravenous blood collection; Device: dCA measurement

INTERVENTIONS:
Device: BB-RIC-D1/LAPUL Medical Devices Co, Ltd, China — The RIC consisted of 4 cycles of extremities ischemia (5-minute blood pressure cuff inflation to 200 mm Hg, followed by 5-minute cuff deflation). The tourniquets were applied to one side upper arm. This intervention was undertaken twice a day for 7 days.
Procedure: Intravenous blood collection — Nurses will collect intravenous blood 3ml four times (at baseline and the first, seventh and eighth day of the study).The blood samples will be stored for laboratory test.The blood samples only use for the trial.
Device: dCA measurement — Serial measurements of dCA were performed at 10 days, baseline, 1st, 2ed, 4th, 7th, 8th, 10th, 14th, 21th and 35th of the study.The continuous ABP was measured non-invasively using a servo-controlled plethysmograph (Finometer Pro, the Netherlands) at the middle finger. Two 2 MHz transcranial Doppler probe was used to measure continuous cerebral blood flow velocity (CBFV) simultaneously in the bilateral middle cerebral arteries at a depth of 45-60 mm Endtidal CO2 was monitored using a capnograph (MultiDop X2, DWL, Sipplingen, Germany). The probes were placed over temporal windows and fixed with a customized head frame. CBFV and continuous arterial blood pressure were recorded simultaneously from each subject in the supine position for 10 minutes. All data were recorded for further assessment and analysis.

SUMMARY:
The purpose of this study is to determine the impact of serial remote ischemic conditioning on dynamic cerebral autoregulation and related hematology indexes in healthy adults.

DETAILED DESCRIPTION:
Remote ischemic conditioning(RIC) is the phenomenon whereby brief cycles of ischemia and reperfusion, applied to a distant organ, provide protection to the target organ. Dynamic cerebral autoregulation(dCA), a mechanism to maintain the cerebral blood flow, has been proved to be critical for the occurrence,development and prognosis of ischemic neurovascular disease. In this study, we hypothesis that RIC provides neuro-protection by means of improving dCA.

ELIGIBILITY:
Inclusion Criteria:

* age from 18 to 50,both genders
* willing to participate in follow-up visits

Exclusion Criteria:

* current or having a history of chronic physical diseases or mental diseases
* suffering from infectious diseases in late one month
* pregnant and lactating women#
* smoking or drinking#
* inability to cooperate sufficiently to complete the dCA examination

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2021-07-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RIC Group
Started | 36
Completed | 22
Not Completed | 14

BASELINE CHARACTERISTICS:
Arm/Group | RIC Group
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.73 (1.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: cm] | 164.50 (8.36)
Weight [Mean (Standard Deviation); unit: kg] | 56.81 (9.42)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 20.88 (2.10)

OUTCOME MEASURES:

1. Primary Outcome: Dynamic Cerebral Autoregulation Parameter: Phase Difference(PD) in Degree
Description: Dynamic cerebral autoregulation (dCA) is an important indicator of cerebrovascular function which related to the prognosis of cerebrovascular disease. DCA is usually calculated by transfer function analysis. Phase Difference (PD) is gengreated. Low PD at a low frequency band indicates impairment of autoregulation, as it suggests that cerebral blood flow velocity follows the changes in arterial blood pressure with a short delay.
Time Frame: 36 days
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | RIC Group
Number analyzed (Participants) | 22
degree | 45.87 (13.02)

2. Secondary Outcome: Dynamic Cerebral Autoregulation Parameter: Gain in cm/s/mmHg
Description: High gain at the same frequency band is also considered an indicator of compromised autoregulation for passively transferring the amplitude of arterial blood pressure to cerebral blood flow velocity.
Time Frame: 36 days
Measure: Mean (Standard Deviation); unit: cm/s/mmHg
Arm/Group | RIC Group
Number analyzed (Participants) | 22
cm/s/mmHg | 0.95 (0.25)

ADVERSE EVENTS:
Time Frame: 36 days
Description: No adverse event was reported.
Arm/Group | RIC Group
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-10): https://cdn.clinicaltrials.gov/large-docs/62/NCT04899362/Prot_SAP_000.pdf